CLINICAL TRIAL: NCT03766243
Title: A Comparison Between Two Educational Methods in the Rehabilitation of the Microstomia in Systemic Sclerosis: a Randomized Controlled Trial
Brief Title: A Comparison Between Two Educational Methods in the Rehabilitation of the Microstomia in Systemic Sclerosis
Acronym: SScM398-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCSS Istituto Dermopatico dell'Immacolata, Fondazione Luigi Maria Monti (Other)
Collaborators: Centro di Eccellenza per la Cultura e la Ricerca Infermieristica (CECRI) (Unknown); Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SScMicrostomia398-1
Record Dates: First submitted 2018-07-19; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Scleroderma, Systemic
Keywords: Microstomia; Rehabilitation; Self-Management
MeSH Terms: conditions — Scleroderma, Systemic; Microstomia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brochure and DVD plus nursing training (Experimental): In addition to the "control intervention", see below, the experimental group was closely followed by the research nurse, an expert in Adult Education, who held 20-minute "face to face" meetings at baseline and at follow-up with the patients allocated to the experimental group. The nurse provided theoretical explanations on the exercises, watched the explanatory DVD with the patients, answering questions and commenting relevant points, and then had the patients repeat the exercises in front of a mirror under direct observation, so that any errors could be pointed out and corrected.
  Interventions: Behavioral: Brochure and DVD plus nursing training
- Brochure and DVD only (Active Comparator): After recruitment, in a 30-minute meeting, a clinical nurse measured the opening of the mouth. She gave each participant the information brochure, the audio-visual DVD for self-management of oral exercises, diary card, and the research questionnaires, and explained their content and use. At the same time, she contacted the research nurse to obtain the random allocation to one of the study groups for that patient.
  These exercises had to be done every day for the entire duration of the program (12 months) and registered in the diary with any comments.
  Interventions: Behavioral: Brochure and DVD only

INTERVENTIONS:
Behavioral: Brochure and DVD plus nursing training — After recruitment for both groups of participants, in a 30-minute meeting, a clinical nurse measured the opening of the mouth. She gave each participant the information brochure, the audio-visual DVD for self-management of oral exercises, diary card, and the research questionnaires, and explained their content and use.
  The intervention consisted of stretching exercises and movements involving the mimic muscles to perform in front of a mirror. The control group could learn the standardized exercises for the mouth-opening through information brochure and the audio-visual DVD.
  The experimental group was closely followed by the research nurse, an expert in Adult Education, who held 20-minute "face to face" meetings at baseline and at follow-up with the patients allocated to the experimental group. For both groups an information brochure and an audio-visual DVD were developed specifically for the study. The audio-visual DVD is available on the IDI-IRCCS institutional website.
  Arms: Brochure and DVD plus nursing training
Behavioral: Brochure and DVD only — After recruitment for both groups of participants, in a 30-minute meeting, a clinical nurse measured the opening of the mouth. She gave each participant the information brochure, the audio-visual DVD for self-management of oral exercises, diary card, and the research questionnaires, and explained their content and use.
  The intervention consisted of stretching exercises and movements involving the mimic muscles to perform in front of a mirror. The control group could learn the standardized exercises for the mouth-opening through information brochure and the audio-visual DVD.
  Arms: Brochure and DVD only

SUMMARY:
Background: A typical feature of SSc is the fibrotic involvement of the connectival tissue of the face, which causes microstomia.

Objectives: To test the effectiveness of an educational intervention with "face to face" training, compared to a standard information program, to reduce microstomia in women with SSc.

Methods: SSc patients were randomized to the experimental and control group. Both groups received written and audiovisual information for self-management of microstomia; in addition, the experimental group received a reinforced training at baseline and at follow-up. Primary outcome: change in inter-incisal distance; secondary outcome: patient-reported mouth disability.

DETAILED DESCRIPTION:
The study was designed as a single-blind, two-arm, randomized controlled study with a 12-month follow-up period. Recruitment started in February 2013 and it continued until January 2015. After recruitment, the patients were seen quarterly (i.e., follow-up visits at 3, 6, 9, and 12 months). Before follow-up visits, patients were contacted by phone to remind them of their appointment.

The participants were inpatients, mainly from Central and Southern Italy, and they were enrolled in a single center, the IDI-IRCCS, FLMM, in Rome, a large dermatological reference center.

Inclusion criteria were diagnosis of Systemic Sclerosis, according to the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) criteria;23 age >18 years; ability to understand the Italian language; subjective perception of problems with opening the mouth, such as hardened tissues, reduced mobility, pain - confirmed by a dermatologist; signed informed consent.

Exclusion criteria were edentulous patients, presence of dental conditions, documented dysfunction of the temporo-mandibular joint, oral neoplasia, sub-mandibular inflammatory conditions, patients already undergoing face massages or face physiotherapy, patients who had undergone mouth lipofilling, patients with severe hand disability (including deep ulcers, and severe pain), and patients with documented psychiatric conditions or taking psychotropic medications.

Randomization The assignment to the intervention and control group was made according to a random sequence generated by a computer program. The randomization list was maintained by an investigator who was not involved in patient recruitment nor in outcome measurement.

Each entry of the randomization list was placed in a sealed envelope, numbered in ascending order, and given to a research nurse after the inclusion/exclusion criteria were verified and the informed consent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SSc, according to the ACR/EULAR criteria;
* age >18 years;
* ability to understand the Italian language;
* subjective perception of problems with opening the mouth, such as hardened tissues, reduced mobility, pain - confirmed by a dermatologist;
* signed informed consent.

Exclusion Criteria:

* edentulous patients,
* presence of dental conditions,
* documented dysfunction of the temporo-mandibular joint,
* oral neoplasia,
* sub-mandibular inflammatory conditions,
* patients already undergoing face massages or face physiotherapy,
* patients who had undergone mouth lipofilling,
* patients with severe hand disability (including deep ulcers, and severe pain),
* patients with documented psychiatric conditions or taking psychotropic medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Interincisal distance | 1 year
  Change in the maximum distance between the tip of the upper and lower incisors, from baseline to 1-year follow-up.

SECONDARY OUTCOMES:
Self-reported severity of mouth disability | 1 year
  To measure mouth disability, the investigators used the Italian version of the standardized self-administered questionnaire Mouth Handicap in Systemic Sclerosis (MHISS). MHISS consists of 12 items (each scored 0-4, with a total score ranging from 0 to 48) divided into 3 subscales: subscale 1 (5 items: 1, 3, 4, 5 and 6; range 0-20) examines handicap related to reduced mouth opening; subscale 2 (5 items: 2, 7, 8, 9 and 10; range 0-20) assesses handicap related to sicca syndrome; and subscale 3 (items 11 and 12; range 0-8) examines aesthetic concerns. The total score is obtained by summing the score for all items. Higher scores denote a greater mouth disability.
Dermatological life quality | 1 year
  Quality of life was measured with the Skindex-17, a dermatology-specific questionnaire consisting of 17 items subdivided into two scales: Symptoms and Psychosocial. Possible range for both scales 0 - 100. Higher scores indicate a greater impact of the disease. Interpretation: for the Symptoms scale, <50 non-severe, >=50 severe; for the Psychosocial scale, <20.82 mild, 20.83-37.50 moderate, >=37.51 severe.
Disease-specific life quality | 1 year
  To measure disease-specific life quality the investigators used the Systemic Sclerosis Questionnaire (SySQ), a self-administered standardized questionnaire whose Italian version was validated in our institution. The SySQ has four scales: General Symptoms, 8 items; Muscle-Skeletal, 11 items; Cardio-Respiratory, 6 items; Gastro-Intestinal, 7 items. Items are all scored 0-3. Scale scores are given by the mean of the items belonging to that scale, again with range 0-3. Higher scores indicate a worse quality of life.
Psychological well-being | 1 year
  Possible presence of anxiety/depression was investigated with a generic questionnaire validated in the field of dermatology, the 12-item General Health Questionnaire-12 (GHQ-12). GHQ-12 items have 4 possible answers, and scores were computed in the conventional way, collapsing adjacent responses to obtain a dichotomous scoring (0 + 0 + 1 + 1). Possible score 0-12. Based on previous research, patients were classified as "GHQ-cases" (i.e., with probable minor non psychotic disorders) if the dichotomous scoring was >=4; and as "GHQ-noncases" if the dichotomous scoring was <4.

CONTACTS AND LOCATIONS:
Overall Officials: Damiano DC Abeni, MD, MPH, Study Chair — IDI-IRCCS, Fondazione Luigi Maria Monti

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naylor WP, Douglass CW, Mix E. The nonsurgical treatment of microstomia in scleroderma: a pilot study. Oral Surg Oral Med Oral Pathol. 1984 May;57(5):508-11. doi: 10.1016/0030-4220(84)90309-8. PMID 6587299
- [Background] Ayala F, de Baranda Andujar PS. Effect of 3 different active stretch durations on hip flexion range of motion. J Strength Cond Res. 2010 Feb;24(2):430-6. doi: 10.1519/JSC.0b013e3181c0674f. PMID 20072058
- [Background] Maddali Bongi S, Del Rosso A, Miniati I, Galluccio F, Landi G, Tai G, Matucci-Cerinic M. The Italian version of the Mouth Handicap in Systemic Sclerosis scale (MHISS) is valid, reliable and useful in assessing oral health-related quality of life (OHRQoL) in systemic sclerosis (SSc) patients. Rheumatol Int. 2012 Sep;32(9):2785-90. doi: 10.1007/s00296-011-2049-x. Epub 2011 Aug 17. PMID 21847653
- [Background] Uras C, Giannantoni P, Tabolli S, DI Giulio P, Peghetti A, Cianchini G, Abeni D. Measuring disability of women with systemic sclerosis: validation of the italian version of the systemic sclerosis questionnaire. G Ital Dermatol Venereol. 2016 Aug;151(4):332-9. Epub 2015 May 13. PMID 25969348
- [Background] Synnot A, Ryan R, Prictor M, Fetherstonhaugh D, Parker B. Audio-visual presentation of information for informed consent for participation in clinical trials. Cochrane Database Syst Rev. 2014 May 9;2014(5):CD003717. doi: 10.1002/14651858.CD003717.pub3. PMID 24809816
- [Background] Kroon FP, van der Burg LR, Buchbinder R, Osborne RH, Johnston RV, Pitt V. Self-management education programmes for osteoarthritis. Cochrane Database Syst Rev. 2014 Jan 15;2014(1):CD008963. doi: 10.1002/14651858.CD008963.pub2. PMID 24425500
- [Background] Lorig K. Partnerships between expert patients and physicians. Lancet. 2002 Mar 9;359(9309):814-5. doi: 10.1016/S0140-6736(02)07959-X. No abstract available. PMID 11897275